CLINICAL TRIAL: NCT04593940
Title: Randomized Master Protocol for Immune Modulators for Treating COVID-19
Brief Title: Immune Modulators for Treating COVID-19
Acronym: ACTIV-1 IM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daniel Benjamin (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Daniel Benjamin, Kiser-Arena Distinguished Professor, Duke University Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00106301
Record Dates: First submitted 2020-09-23; First posted 2020-10-20 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Covid19
Keywords: COVID19
MeSH Terms: conditions — COVID-19 | interventions — Infliximab; Abatacept; remdesivir; cenicriviroc

STUDY DESIGN:
Intervention Model Description: ACTIV-1 IM builds upon findings and the model used for other network COVID studies. Including multiple therapeutic agents under a single protocol avoids duplication of effort in terms of infrastructure, trial governance, information systems (EDC, web-based randomization, etc.) and other aspects of study management. Implementation of the master protocol facilitates discontinuation of less promising agents and addition of possibly newly emergent agents that become available after the study begins, without stopping and starting the study itself for extended pauses.
  All test agents are evaluated as add-on therapies to the local SoC at each clinic. The master protocol design allows for the efficacy and safety of each agent to be determined based on comparisons with a pooled control group, consisting of patients receiving SoC plus placebo. Sharing control patients across all test agents substantially reduces the sample size requirements for the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study Drug and Matching Placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Standard of Care + infliximab or matching placebo (Active Comparator): infliximab (single dose IV 5mg/kg given on day 1) or matching placebo
  Interventions: Drug: Infliximab; Drug: Remdesivir
- Standard of Care + abatacept or matching placebo (Active Comparator): abatacept (single dose IV 10 mg/kg up to 1,000 mg given on day 1) or matching placebo
  Interventions: Drug: Abatacept; Drug: Remdesivir
- Standard of Care + cenicriviroc or matching placebo (closed to enrollment as of 3-Sep-2021) (Active Comparator): cenicriviroc [tablet, Day 1/Loading Dose: 450 mg (300mg morning and 150mg evening) Day 2 - 29/Maintenance Dose: 300 mg (150 mg BID) through Day 29]. or matching placebo
  Interventions: Drug: Remdesivir; Drug: cenicriviroc (closed to enrollment as of 3-Sep-2021)

INTERVENTIONS:
Drug: Infliximab — study drug or matching placebo
  Other Names: remicade
  Arms: Standard of Care + infliximab or matching placebo
Drug: Abatacept — study drug or matching placebo
  Other Names: orencia
  Arms: Standard of Care + abatacept or matching placebo
Drug: Remdesivir — Standard of Care
Drug: cenicriviroc (closed to enrollment as of 3-Sep-2021) — study drug or matching placebo
  Arms: Standard of Care + cenicriviroc or matching placebo (closed to enrollment as of 3-Sep-2021)

SUMMARY:
ACTIV-1 IM is a master protocol designed to evaluate multiple investigational agents for the treatment of moderately or severely ill patients infected with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The research objectives are to evaluate each agent with respect to speed of recovery, mortality, illness severity, and hospital resource utilization. Each agent will be evaluated as add-on therapy to the standard of care (SoC) in use at the local clinics, including remdesivir (provided). The SoC may change during the course of the study based on other research findings. Comparisons of the agents among themselves is not a research objective.

The study population corresponds to moderately and severely ill patients infected with the coronavirus disease 2019 (COVID-19) virus. Recruitment will target patients already hospitalized for treatment of COVID-19 infection as well as patients being treated for COVID-19 infection in Emergency Departments while waiting to be admitted to the hospital. Patients both in and out of the ICU are included in the study population.

DETAILED DESCRIPTION:
ACTIV-1 IM is a master protocol designed to evaluate immune modulators for the treatment of moderately or severely ill hospitalized patients infected with COVID-19. Trial participants will be assessed daily while hospitalized. If the participants are discharged from the hospital prior to Day 29, they will have follow-up study visits at Days 8, 11, 15, 22, and 29. For discharged participants, it is preferred that the Day 8, 11, 15, and 29 visits are in person to obtain safety laboratory tests and blood (serum/plasma) samples for secondary research as well as clinical outcome data. However, infection control or other restrictions may limit the ability of the participant to return to the clinic. In this case, these visits may be conducted by phone, and only clinical data will be obtained. The Day 22 visit does not have laboratory tests or collection of samples and is conducted by phone. The Day 60 assessment will be conducted by phone.

The effectiveness of each therapeutic agent as add-on therapy to SoC plus remdesivir (provided) will be evaluated based on the primary endpoint of time to recovery by Day 29. The sample size requirements are based on the ability to detect a moderate improvement in time to recovery (3-4 fewer days) for each agent. A total of 788 recoveries are required for each comparison to provide approximately 85% power to detect a recovery rate ratio of 1.25. Assuming 73% of participants achieve recovery in 28 days, consistent with the ACTT-1 results, the total sample size to evaluate 1, 2, and 3 agents in ACTIV-1 IM is approximately 1080, 1620, and 2160, respectively. Because each agent is being compared to SoC with no between-agent comparisons, no multiplicity adjustments for multiple agents are planned.

The CVC arm of the study was closed to enrollment on 3-Sep-2021.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to a hospital or awaiting admission in the ED with symptoms suggestive of COVID-19.
2. Subject (or legally authorized representative) provides informed consent prior to initiation of any study procedures.
3. Subject (or legally authorized representative) understands and agrees to comply with planned study procedures.
4. Male or non-pregnant female adults ≥18 years of age at time of enrollment.
5. Has laboratory-confirmed (within 14 days prior to enrollment) SARS-CoV-2 infection as determined by PCR or other commercial or public health assay in any specimen.
6. Ongoing illness of any duration, and at least one of the following:

   * Radiographic infiltrates by imaging (chest x-ray, CT scan, etc.), OR
   * Blood oxygen saturation (SpO2) ≤94% on room air, OR
   * Requiring supplemental oxygen, OR
   * Requiring mechanical ventilation or ECMO.
7. Women of childbearing potential must agree to either abstinence or use of at least one primary form of contraception not including hormonal contraception from the time of screening through Day 60.
8. Agrees to not to participate in another interventional trial for the treatment of COVID-19 through Day 60.

Exception 1: Participant may co-enroll in ACTIV-4 (ACTIV-4A and ACTIV-4C). Exception 2: Participants in ACTIV-2 who have been hospitalized may be enrolled in ACTIV-1 as long as ACTIV-2 study therapy has been discontinued. They will remain in ACTIV-2 follow-up.

Exception 3: If participant is already participating in a COVID-19 vaccine trial but develops COVID-19 disease that requires hospitalization, participant is eligible for this study, assuming all other inclusion/exclusion criteria are met.

Exclusion Criteria:

1. ALT or AST >10 times the upper limit of normal.
2. Estimated glomerular filtration rate (eGFR) <30 mL/min (including patients receiving hemodialysis or hemofiltration).

   Exception: Participants with an eGFR <30 mL/min may enroll as long as their renal insufficiency has been stable without renal replacement therapy for ≥1 month and they are not current candidates for renal replacement therapy. These participants will not receive remdesivir.
3. Neutropenia (absolute neutrophil count <1000 cells/μL) (<1.0 x 103/μL or <1.0 GI/L).
4. Lymphopenia (absolute lymphocyte count <200 cells/μL) (<0.20 x 103/μL or <0.20 GI/L)
5. Pregnancy or breast feeding.
6. Anticipated discharge from the hospital or transfer to another hospital which is not a study site within 72 hours.
7. Known allergy to any study medication.
8. Received cytotoxic or biologictargeted immune-modulator treatments (such as anti-interleukin-1 [IL-1], anti-IL-6 [tocilizumab or sarilumab], anti-IL-17, or T-cell or B-cell targeted therapies ([e.g., rituximab), tyrosine kinase], JAK inhibitors [including baricitinib,], TNF inhibitors, or interferon) within 4 weeks or 5 half-lives prior to screening., whichever is longer. Steroid dependency, defined as need for prednisone at a dose >10 mg (or equivalent) for >1 month within 2 weeks of screening, is exclusionary. Note Exception 1: Dexamethasone (at a dose of 6 mg per day for up to 10 days) is permitted for the treatment of COVID-19 in patients who are already mechanically ventilated and in patients who require supplemental oxygen at screening, but who are not mechanically ventilated in accordance with national guidelines. Note Exception 2: Infusion of convalescent plasma given for treatment of COVID-19 while on-study is also allowed.

   Exception 3: Monoclonal antibody therapy given for COVID-19 treatment at any time prior to enrollment is also allowed.
9. BasedKnown or suspected history of untreated tuberculosis (TB). TB diagnosis may be suspected based on medical history and concomitant therapies that would suggest TB infection, have suspected clinical diagnosis of current active tuberculosis (TB) or, if. Participants are also excluded if they have known, latent TB treated for less than 4 weeks with appropriate anti-tuberculosis therapy per local guidelines (by history only, no screening required).
10. Based on medical history and concomitant therapies that would suggest infection,Known or suspected serious, active bacterial, fungal, or viral (infection (excepting SARS-CoV-2 and including, but not limited to, active HBV, HCV, or HIV/AIDS). with the latter defined as a CD4 count <200 or an unsuppressed HIV viral load), or other infection (besides COVID-19) that in the opinion of the investigator could constitute a risk when taking investigational product.

    Note: Broad-spectrum empiric antibiotic usage does not exclude participation.
11. Have received any live vaccine (that is,or live attenuated) within 3 months before screening, or intend to receive a live vaccine (or live attenuated) during the study. Note Exception: Use of prior non-live (inactivated) vaccinations is allowed for all participants, including any vaccine for COVID-19.
12. Severe hepatic impairment (defined as liver cirrhosis Child stage C).
13. CurrentKnown severe heart failure (New York Heart Association [NYHA] III-IV).) or new-onset left-systolic or global cardiac dysfunction in the setting of COVID-19.

    Exception: Right-sided heart dysfunction or pulmonary hypertension thought related to COVID-19 is permitted.
14. In the Investigator's judgment, the patient has any advanced organ dysfunction that would not make participation appropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1971 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel K Benjamin, MD, PhD, Principal Investigator — Duke University; Bill Powderly, MD, Study Chair — Washington University School of Medicine
Locations (91):
- United States (67):
  - Banner University Medical Center, Phoenix, Arizona
  - University of Arkansas Medical Sciences, Little Rock, Arkansas
  - Scripps Clinical Medical Group, La Jolla, California
  - UCLA - Ronald Reagan Medical Center, Los Angeles, California
  - Riverside University, Moreno Valley, California
  - UC Irvine Medical Center, Orange, California
  - Stanford University Medical Center, Palo Alto, California
  - UCLA Medical Center- Santa Monica, Santa Monica, California
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida-Jacksonville, Jacksonville, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Tulane School of Medicine, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - U Mass Memorial Medical Center, Worcester, Massachusetts
  - U Mass University Medical Center, Worcester, Massachusetts
  - MidMichigan Medical Center- Gratiot, Alma, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Health Care, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Trinitas Hospital, Elizabeth, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers New Jersey Medical School, New Brunswick, New Jersey
  - NYU Brooklyn, Brooklyn, New York
  - University at Buffalo, Buffalo, New York
  - Flushing Hospital Medical Center, Flushing, New York
  - Jamaica Hospital Medical Center, Jamaica, New York
  - NYU Long Island, Long Island City, New York
  - New York University Langone Medical Center, New York, New York
  - Harlem Hospital Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - St Lawrence Health System, Potsdam, New York
  - University of Rochester Medical Center-Strong Memorial Hospital, Rochester, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Mercy Saint Vincent Medical Center, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Reading Hospital Study, Wyomissing, Pennsylvania
  - Avera McKennan Hospital, Sioux Falls, South Dakota
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Methodist Health System Clinical Research Institute, Dallas, Texas
  - University of Texas Health Science Center - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Trinity Mother Frances Hospital, Tyler, Texas
  - University of Texas Health Center at Tyler, Tyler, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Providence Medical Research Center, Spokane, Washington
  - West Virginia University, Morgantown, West Virginia
  - Gundersen Health System, La Crosse, Wisconsin
- Argentina (9):
  - Hospital Interzonal Dr Jose Penna Bahia Blanca, Bahía Blanca, Buenos Aires
  - Sanatorio Ramon Cereijo, CABA, Buenos Aires
  - Instituto Medico Platense, La Plata, Buenos Aires
  - Clinica Central S.A., Villa Regina, Río Negro Province
  - Hospital Ramos Mejia, Buenos Aires
  - Hospital Rawson, Córdoba
  - Sanatorio Allende, Córdoba
  - Sanatorio Britanico, Rosario
  - Sanatorio Diagnóstico/ Instituto del Buen Aire, Santa Fe
- Brazil (7):
  - Hospital Brasília, Brasília, Federal District
  - Hospital Felício Rocho, Belo Horizonte, Minas Gerais
  - Instituto DOR de Ensino e Pesquisa Hospital Glória D'Or, Rio de Janeiro, Rio de Janeiro / RJ
  - Hospital Ernesto Dornelles, Porto Alegre, Rio Grande D Sul /RS
  - Hospital de Clinicas de Porto Alegre HCPA, Porto Alegre, Rio Grande Do Sul / RS
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande Do Sul/RS
  - Hospital e Maternidade Celso Pierro - PUC Campinas, Campinas, São Paulo/SP
- Mexico (2):
  - Nuevo Hospital Civil de Guadalajara "Dr. Juan I. Menchaca", Guadalajara, Guadalajara Jalisco
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Nuevo León, Monterrey
- Peru (6):
  - Hospital Central FAP, Lima, Lima/Lima
  - Hospital Regional Lambayeque, Chiclayo
  - Hospitala Nacional Hipólito Unánue, Lima
  - Hospital Nacional Aezobispo Loayza, Lima
  - Hospital de Chancay y Servicios Basicos de Salud, Lima
  - Clínica Belén SANNA, Piura

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lachiewicz AM, Shah M, Der T, Cyr D, Al-Khalidi HR, Lindsell C, Iyer V, Khan A, Panettieri R, Rauseo AM, Maillo M, Schmid A, Jagpal S, Powderly WG, Bozzette SA; ACTIV-1 IM study group members. Resource Use in the Randomized Master Protocol for Immune Modulators for Treating COVID-19 (ACTIV-1 IM): A Secondary Data Analysis. CHEST Crit Care. 2024 Dec;2(4):100095. doi: 10.1016/j.chstcc.2024.100095. Epub 2024 Aug 22. PMID 39610848
- [Derived] Balevic SJ, Benjamin DK Jr, Powderly WG, Smith PB, Gonzalez D, McCarthy MW, Shaw LK, Lindsell CJ, Bozzette S, Williams D, Linas BP, Blamoun J, Javeri H, Hornik CP; ACTIV-1 IM Study Group. Abatacept Pharmacokinetics and Exposure Response in Patients Hospitalized With COVID-19: A Secondary Analysis of the ACTIV-1 IM Randomized Clinical Trial. JAMA Netw Open. 2024 Apr 1;7(4):e247615. doi: 10.1001/jamanetworkopen.2024.7615. PMID 38662372
- [Derived] O'Halloran JA, Ko ER, Anstrom KJ, Kedar E, McCarthy MW, Panettieri RA Jr, Maillo M, Nunez PS, Lachiewicz AM, Gonzalez C, Smith PB, de Tai SM, Khan A, Lora AJM, Salathe M, Capo G, Gonzalez DR, Patterson TF, Palma C, Ariza H, Lima MP, Blamoun J, Nannini EC, Sprinz E, Mykietiuk A, Alicic R, Rauseo AM, Wolfe CR, Witting B, Wang JP, Parra-Rodriguez L, Der T, Willsey K, Wen J, Silverstein A, O'Brien SM, Al-Khalidi HR, Maldonado MA, Melsheimer R, Ferguson WG, McNulty SE, Zakroysky P, Halabi S, Benjamin DK Jr, Butler S, Atkinson JC, Adam SJ, Chang S, LaVange L, Proschan M, Bozzette SA, Powderly WG; ACTIV-1 IM Study Group Members. Abatacept, Cenicriviroc, or Infliximab for Treatment of Adults Hospitalized With COVID-19 Pneumonia: A Randomized Clinical Trial. JAMA. 2023 Jul 25;330(4):328-339. doi: 10.1001/jama.2023.11043. PMID 37428480
- [Derived] Ko ER, Anstrom KJ, Panettieri RA, Lachiewicz AM, Maillo M, O'Halloran JA, Boucher C, Smith PB, McCarthy MW, Segura Nunez P, Mendivil Tuchia de Tai S, Khan A, Mena Lora AJ, Salathe M, Kedar E, Capo G, Rodriguez Gonzalez D, Patterson TF, Palma C, Ariza H, Patelli Lima M, Blamoun J, Nannini EC, Sprinz E, Mykietiuk A, Wang JP, Parra-Rodriguez L, Der T, Willsey K, Benjamin DK, Wen J, Zakroysky P, Halabi S, Silverstein A, McNulty SE, O'Brien SM, Al-Khalidi HR, Butler S, Atkinson J, Adam SJ, Chang S, Maldonado MA, Proscham M, LaVange L, Bozzette SA, Powderly WG; ACTIV-1 IM study group members. Abatacept for Treatment of Adults Hospitalized with Moderate or Severe Covid-19. medRxiv [Preprint]. 2022 Sep 26:2022.09.22.22280247. doi: 10.1101/2022.09.22.22280247. PMID 36203544
- [Derived] O'Halloran JA, Kedar E, Anstrom KJ, McCarthy MW, Ko ER, Nunez PS, Boucher C, Smith PB, Panettieri RA, de Tai SMT, Maillo M, Khan A, Mena Lora AJ, Salathe M, Capo G, Gonzalez DR, Patterson TF, Palma C, Ariza H, Lima MP, Lachiewicz AM, Blamoun J, Nannini EC, Sprinz E, Mykietiuk A, Alicic R, Rauseo AM, Wolfe CR, Witting B, Benjamin DK, McNulty SE, Zakroysky P, Halabi S, Butler S, Atkinson J, Adam SJ, Melsheimer R, Chang S, LaVange L, Proschan M, Bozzette SA, Powderly WG; ACTIV-1 IM study group members. Infliximab for Treatment of Adults Hospitalized with Moderate or Severe Covid-19. medRxiv [Preprint]. 2022 Sep 26:2022.09.22.22280245. doi: 10.1101/2022.09.22.22280245. PMID 36172138
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care + Infliximab: infliximab (single dose IV 5mg/kg given on day 1)
  Infliximab: study drug Remdesivir: Standard of Care
- Standard of Care + Abatacept: abatacept (single dose IV 10 mg/kg up to 1,000 mg given on day 1)
  Abatacept: study drug
  Remdesivir: Standard of Care
- Standard of Care + Cenicriviroc: cenicriviroc [tablet, Day 1/Loading Dose: 450 mg (300mg morning and 150mg evening) Day 2 - 29/Maintenance Dose: 300 mg (150 mg BID) through Day 29].
  Remdesivir: Standard of Care
  cenicriviroc (closed to enrollment as of 3-Sep-2021): study drug
- Shared Placebo: Shared placebo
  Placebo group was shared among up to all 3 arms for which the participant qualified.
Period: Overall Study
Arm/Group | Standard of Care + Infliximab | Standard of Care + Abatacept | Standard of Care + Cenicriviroc | Shared Placebo
Started | 531 | 524 | 360 | 556
Completed | 425 | 394 | 263 | 419
Not Completed | 106 | 130 | 97 | 137

BASELINE CHARACTERISTICS:
Groups:
- Shared Placebo: placebo group
  placebo group was shared among up to all 3 arms; whichever arms the participant qualified.
- Total: Total of all reporting groups
Arm/Group | Standard of Care + Infliximab | Standard of Care + Abatacept | Standard of Care + Cenicriviroc | Shared Placebo | Total
Number analyzed (Participants) | 531 | 524 | 360 | 556 | 1971
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (14.87) | 54.8 (14.65) | 54.7 (14.32) | 55.0 (14.66) | 54.8 (14.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 198 | 197 | 123 | 235 | 753
  Male | 333 | 327 | 237 | 321 | 1218
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 257 | 219 | 159 | 270 | 905
  Not Hispanic or Latino | 264 | 283 | 187 | 275 | 1009
  Unknown or Not Reported | 10 | 22 | 14 | 11 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 5 | 4 | 5 | 19
  Asian | 12 | 16 | 11 | 17 | 56
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 0 | 2
  Black or African American | 80 | 74 | 44 | 76 | 274
  White | 328 | 325 | 226 | 350 | 1229
  More than one race | 2 | 0 | 2 | 3 | 7
  Unknown or Not Reported | 103 | 103 | 73 | 105 | 384
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 56 | 52 | 33 | 64 | 205
  United States | 344 | 352 | 241 | 354 | 1291
  Brazil | 54 | 46 | 38 | 57 | 195
  Mexico | 15 | 18 | 8 | 18 | 59
  Peru | 62 | 56 | 40 | 63 | 221

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Recovered by Day 28
Description: Time to recovery by day 28. The number of participants who have recovered by day 28.
Time Frame: Days 1-28
Population: Intent to treat population. This study had a shared placebo group meaning some participants are included in the analysis for multiple placebo comparison groups. Per master protocol design patients randomized to placebo had the potential to be included in the analyses for infliximab, abatacept, and cenicriviroc based on their eligibility. Therefore, the counts of participants will be higher than the number of participants enrolled.
Measure: Count of Participants; unit: Participants
Groups:
- Standard of Care + Infliximab Matching Placebo: infliximab placebo (single dose IV 5mg/kg given on day 1)
  Remdesivir: Standard of Care
- Standard of Care + Abatacept Matching Placebo: abatacept matching placebo(single dose IV 10 mg/kg up to 1,000 mg given on day 1)
  Remdesivir: Standard of Care
- Standard of Care + Cenicriviroc: cenicriviroc [tablet, Day 1/Loading Dose: 450 mg (300mg morning and 150mg evening) Day 2 - 29/Maintenance Dose: 300 mg (150 mg BID) through Day 29].
  Remdesivir: Standard of Care
  cenicriviroc or matching placebo arm closed to enrollment as of 3-Sep-2021
- Standard of Care + Cenicriviroc Matching Placebo: cenicriviroc matching placebo [tablet, Day 1:Loading Dose: 450 mg (300mg morning and 150mg evening) Day 2 - 29/Maintenance Dose: 300 mg (150 mg BID) through Day 29].
  Remdesivir: Standard of Care
  cenicriviroc or matching placebo arm closed to enrollment as of 3-Sep-2021
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 531 | 530 | 524 | 525 | 360 | 363
Participants | 421 | 405 | 414 | 397 | 273 | 287
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; p = 0.0793, Fine-Gray Proportional Hazards Model; Recovery Rate Ratio = 1.122, 95% CI 2-sided [0.987 to 1.275]
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; p = 0.0864, Fine-Gray Proportional Hazards Model; Recovery Rate Ratio = 1.120, 95% CI 2-sided [.984 to 1.275]
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; p = 0.9354, Fine-Gray Proportional Hazards Model; Recovery Rate Ratio = 1.006, 95% CI 2-sided [0.862 to 1.176]

2. Secondary Outcome: Number of Participants With Clinical Status for Day 14 Using an 8 Point Ordinal Scale
Description: 8-point ordinal scale assessing clinical status (1=Death is worst, 8=not hospitalized/no limitations on activities is best) To determine a participant's clinical status using the ordinal scale their clinical status was collected at Day 15 assessing day 14.
  The scale used in this study is as follows (from worst to best):
  1. Death;
  2. Hospitalized, on invasive mechanical ventilation or ECMO;
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical in-patient care (COVID-19 related or otherwise);
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical in-patient care; This would include those kept in hospital for quarantine/infection control/social reasons, awaiting bed in rehabilitation facility or homecare, etc.
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized,
Time Frame: Day 14
Population: Intention to treat. This study had a shared placebo group meaning some participants are included in the analysis for multiple placebo comparison groups. Missing data: Infliximab arms 49, Abatacept arms 57, CVC arms 27. Per master protocol design patients randomized to placebo had the potential to be included in the analyses for infliximab, abatacept, and cenicriviroc based on their eligibility. Therefore, the counts of participants will be higher than the number of participants enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 506 | 506 | 493 | 499 | 350 | 346
Participants
  1-Death | 29 | 42 | 24 | 40 | 31 | 25
  2-Hospitalized, on invasive mechanical ventilation or ECMO | 60 | 65 | 63 | 66 | 41 | 38
  3-Hospitalized, on non-invasive ventilation or high flow oxygen devices | 19 | 23 | 31 | 26 | 17 | 15
  4-Hospitalized, requiring supplemental oxygen | 44 | 34 | 38 | 34 | 22 | 29
  5-Hospitalized, not requiring supplemental oxygen - requiring ongoing medical in-patient care | 4 | 11 | 13 | 11 | 6 | 10
  6-Hospitalized, not requiring supplemental oxygen - no longer requires in-patient care | 2 | 2 | 0 | 2 | 1 | 1
  7-Not hospitalized, limitation on activities and/or requiring home oxygen | 163 | 174 | 174 | 173 | 134 | 130
  8-Not hospitalized | 185 | 155 | 150 | 147 | 98 | 98
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; p = 0.0213, Regression, Logistic; Ordinal logistic regression; Odds Ratio (OR) = 1.309, 95% CI 2-sided [1.041 to 1.647] — Ordinal logistic regression
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; p = 0.1732, Regression, Logistic; Ordinal logistic regression; Odds Ratio (OR) = 1.174, 95% CI 2-sided [0.932 to 1.480] — Ordinal logistic regression
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; p = 0.6823, Regression, Logistic; Ordinal logistic regression; Odds Ratio (OR) = 0.944, 95% CI 2-sided [0.717 to 1.243] — Ordinal logistic regression

3. Secondary Outcome: Mortality Through 28 Days
Description: mortality at day 28
Time Frame: Day 1-28
Population: Intent to treat. This study had a shared placebo group meaning some participants are included in the analysis for multiple placebo comparison groups. Per master protocol design patients randomized to placebo had the potential to be included in the analyses for infliximab, abatacept, and cenicriviroc based on their eligibility. Therefore, the counts of participants will be higher than the number of participants enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 531 | 530 | 524 | 525 | 360 | 363
Participants | 53 | 75 | 56 | 77 | 49 | 42
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; p = 0.0229, Regression, Logistic; Odds Ratio (OR) = 0.614, 95% CI 2-sided [0.403 to 0.935]
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; p = 0.0281, Regression, Logistic; Odds Ratio (OR) = 0.629, 95% CI 2-sided [0.416 to 0.951]
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; p = 0.541, Regression, Logistic; Odds Ratio (OR) = 1.167, 95% CI 2-sided [0.711 to 1.917]

4. Secondary Outcome: Number of Participants With Clinical Status for Day 28 Using an 8 Point Ordinal Scale
Description: 8-point ordinal scale assessing clinical status (1=Death is worst, 8=not hospitalized/no limitations on activities is best) To determine a participant's clinical status using the ordinal scale their clinical status was collected at Day 29 assessing day 28.
  The scale used in this study is as follows (from worst to best):
  1. Death;
  2. Hospitalized, on invasive mechanical ventilation or ECMO;
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical in-patient care (COVID-19 related or otherwise);
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical in-patient care; This would include those kept in hospital for quarantine/infection control/social reasons, awaiting bed in rehabilitation facility or homecare, etc.
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized,
Time Frame: Day 28
Population: Intent to treat. This study had a shared placebo group meaning some participants are included in the analysis for multiple placebo comparison groups. Per master protocol design patients randomized to placebo had the potential to be included in the analyses for infliximab, abatacept, and cenicriviroc based on their eligibility. Therefore, the counts of participants will be higher than the number of participants enrolled. Missing data: Infliximab arms 65, Abatacept arms 69, CVC arms 41.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 496 | 500 | 487 | 493 | 338 | 344
Participants
  1-Death | 53 | 75 | 56 | 77 | 49 | 42
  2-Hospitalized, on invasive mechanical ventilation or ECMO | 28 | 27 | 27 | 26 | 25 | 19
  3-Hospitalized, on non-invasive ventilation or high flow oxygen devices | 6 | 7 | 5 | 8 | 7 | 5
  4-Hospitalized, requiring supplemental oxygen | 11 | 10 | 10 | 12 | 4 | 8
  5-Hospitalized, not requiring supplemental oxygen - requiring ongoing medical in-patient care | 3 | 6 | 8 | 5 | 2 | 4
  6-Hospitalized, not requiring supplemental oxygen - no longer requires in-patient care | 2 | 2 | 1 | 2 | 0 | 2
  7-Not hospitalized, limitation on activities and/or requiring home oxygen | 135 | 156 | 149 | 156 | 109 | 115
  8-Not hospitalized | 258 | 217 | 231 | 207 | 142 | 149
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; p = 0.0032, Regression, Logistic; Ordinal logistic regression; Odds Ratio (OR) = 1.435, 95% CI 2-sided [1.129 to 1.825] — Ordinal logistic regression
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; p = 0.0228, Regression, Logistic; Ordinal logistic regression; Odds Ratio (OR) = 1.338, 95% CI 2-sided [1.041 to 1.718] — Ordinal logistic regression
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; p = 0.4994, Regression, Logistic; Ordinal logistic regression; Odds Ratio (OR) = 0.904, 95% CI 2-sided [0.675 to 1.211] — Ordinal logistic regression

5. Secondary Outcome: Mortality Through 14 Days
Description: mortality at day 14
Time Frame: Day 1-14
Population: Intention to treat. This study had a shared placebo group meaning some participants are included in the analysis for multiple placebo comparison groups. Per master protocol design patients randomized to placebo had the potential to be included in the analyses for infliximab, abatacept, and cenicriviroc based on their eligibility. Therefore, the counts of participants will be higher than the number of participants enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 531 | 530 | 524 | 525 | 360 | 363
Participants | 29 | 42 | 24 | 40 | 31 | 25
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; p = 0.0988, Regression, Logistic; Ordinal logistic regression; Odds Ratio (OR) = 0.632, 95% CI 2-sided [0.367 to 1.090] — Ordinal logistic regression
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; p = 0.0354, Regression, Logistic; Ordinal logistic regression; Odds Ratio (OR) = 0.552, 95% CI 2-sided [0.317 to 0.960] — Ordinal logistic regression
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; p = 0.4132, Regression, Logistic; Ordinal logistic regression; Odds Ratio (OR) = 1.287, 95% CI 2-sided [0.703 to 2.355] — Ordinal logistic regression

6. Secondary Outcome: Number of Participants Who Met a One Point Improvement in One Category From Day 0 (Baseline) to Day 28 Using an 8-point Ordinal Scale
Description: 8-point ordinal scale assessing clinical status (1=Death is worst, 8=not hospitalized/no limitations on activities is best). Number of people who met a 1 point improvement.
  The scale used in this study is as follows (from worst to best):
  1. Death;
  2. Hospitalized, on invasive mechanical ventilation or ECMO;
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical in-patient care (COVID-19 related or otherwise);
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical in-patient care; This would include those kept in hospital for quarantine/infection control/social reasons, awaiting bed in rehabilitation facility or homecare, etc.
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized, no limitations on activities.
Time Frame: Day 1-day 28
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 531 | 530 | 524 | 525 | 360 | 363
Participants | 446 | 429 | 435 | 421 | 287 | 302
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; p = 0.1601, Fine-Gray Proportional Hazards Model; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [1.00 to 1.28]
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; p = 0.3550, Fine-Gray Proportional Hazards Model; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.97 to 1.24]
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; p = 0.2386, Fine-Gray Proportional Hazards Model; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.80 to 1.07]

7. Secondary Outcome: Number of Participants Who Met a One Point Improvement in Two Categories From Day 0 (Baseline) to Day 28 Using an 8-point Ordinal Scale
Description: 8-point ordinal scale assessing clinical status (1=Death is worst, 8=not hospitalized/no limitations on activities is best). Number of people who met a two category improvement.
  The scale used in this study is as follows (from worst to best):
  1. Death;
  2. Hospitalized, on invasive mechanical ventilation or ECMO;
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical in-patient care (COVID-19 related or otherwise);
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical in-patient care; This would include those kept in hospital for quarantine/infection control/social reasons, awaiting bed in rehabilitation facility or homecare, etc.
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized, no limitations on activities.
Time Frame: Day 1- day 28
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 531 | 530 | 524 | 525 | 360 | 363
Participants | 429 | 415 | 421 | 406 | 282 | 292
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; p = 0.1519, Fine-Gray Proportional Hazards Model; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.98 to 1.26]
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; p = 0.2605, Fine-Gray Proportional Hazards Model; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.98 to 1.26]
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; p = 0.4359, Fine-Gray Proportional Hazards Model; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.83 to 1.13]

8. Secondary Outcome: Mean Change in the 8-point Ordinal Scale From Day 0 to Day 2
Description: 8-point ordinal scale assessing clinical status (1=Death is worst, 8=not hospitalized/no limitations on activities is best)
Time Frame: Day 0 to day 2
Population: Intent to treat. This study had a shared placebo group meaning some participants are included in the analysis for multiple placebo comparison groups. Per master protocol design patients randomized to placebo had the potential to be included in the analyses for infliximab, abatacept, and cenicriviroc based on their eligibility. Therefore, the counts of participants will be higher than the number of participants enrolled. Missing data: Infliximab arms 24, Abatacept arms 22, CVC arms 9.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 519 | 522 | 512 | 515 | 356 | 358
units on a scale | 3.5 (0.9104) | 3.5 (1.0515) | 3.6 (1.0973) | 3.5 (1.0403) | 3.5 (0.9914) | 3.5 (1.0118)
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; p = 0.3210, t-test, 2 sided; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.18 to 0.06]
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; p = 0.5275, t-test, 2 sided; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.09 to 0.17]
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; p = 0.9993, t-test, 2 sided; Mean Difference (Net) = 0.00, 95% CI 2-sided [-0.15 to 0.15]

9. Secondary Outcome: Mean Change in the 8-point Ordinal Scale From Day 0 to Day 4
Description: 8 point ordinal scale assessing clinical status (1=death is worst, 8=not hospitalized/no limitations on activities is best)
Time Frame: Day 0 to day 4
Population: Intent to treat. This study had a shared placebo group meaning some participants are included in the analysis for multiple placebo comparison groups. Per master protocol design patients randomized to placebo had the potential to be included in the analyses for infliximab, abatacept, and cenicriviroc based on their eligibility. Therefore, the counts of participants will be higher than the number of participants enrolled.Missing data: Infliximab arms 25, Abatacept arms 32, CVC arms 16.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 519 | 517 | 507 | 510 | 352 | 355
units on a scale | 3.9 (1.6004) | 3.9 (1.5320) | 4.0 (1.6526) | 3.9 (1.5468) | 3.9 (1.6385) | 3.9 (1.5624)
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; p = 0.4982, t-test, 2 sided; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.13 to 0.26]
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; p = 0.3491, t-test, 2 sided; Mean Difference (Net) = 0.09, 95% CI 2-sided [-0.10 to 0.29]
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; p = 0.9020, t-test, 2 sided; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.25 to 0.22]

10. Secondary Outcome: Mean Change in the 8-point Ordinal Scale From Day 0 to Day 7
Description: 8-point ordinal scale assessing clinical status (1=death is worst, 8=not hospitalized/no limitations on activities=best)
Time Frame: Day 0 to day 7
Population: Intent to treat. This study had a shared placebo group meaning some participants are included in the analysis for multiple placebo comparison groups. Per master protocol design patients randomized to placebo had the potential to be included in the analyses for infliximab, abatacept, and cenicriviroc based on their eligibility. Therefore, the counts of participants will be higher than the number of participants enrolled.Missing data: Infliximab arms 35, Abatacept arms 43, CVC arms 19.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 514 | 512 | 501 | 505 | 352 | 352
units on a scale | 5.0 (2.2738) | 4.8 (2.2470) | 4.9 (2.2261) | 4.8 (2.2585) | 4.8 (2.2636) | 4.9 (2.2475)
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; p = 0.0842, t-test, 2 sided; Mean Difference (Net) = 0.24, 95% CI 2-sided [-0.03 to 0.52]
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; p = 0.5328, t-test, 2 sided; Mean Difference (Net) = 0.09, 95% CI 2-sided [-0.19 to 0.37]
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; p = 0.4727, t-test, 2 sided; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.46 to 0.21]

11. Secondary Outcome: Mean Change in the 8-point Ordinal Scale From Day 0 to Day 10
Description: as for outcome 8
Time Frame: Day 0 to day 10
Population: Intent to treat. This study had a shared placebo group meaning some participants are included in the analysis for multiple placebo comparison groups. Per master protocol design patients randomized to placebo had the potential to be included in the analyses for infliximab, abatacept, and cenicriviroc based on their eligibility. Therefore, the counts of participants will be higher than the number of participants enrolled. Missing data: Infliximab arms 45, Abatacept arms 51, CVC arms 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 509 | 507 | 498 | 500 | 351 | 348
units on a scale | 5.6 (2.3910) | 5.3 (2.4308) | 5.4 (2.3310) | 5.3 (2.4306) | 5.3 (2.4493) | 5.3 (2.3746)
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; p = 0.0399, t-test, 2 sided; Mean Difference (Net) = 0.31, 95% CI 2-sided [0.01 to 0.61]
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; p = 0.4515, t-test, 2 sided; Mean Difference (Net) = 0.11, 95% CI 2-sided [-0.18 to 0.41]
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; p = 0.6960, t-test, 2 sided; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.43 to 0.29]

12. Secondary Outcome: Mean Change in the 8-point Ordinal Scale From Day 0 to Day 14
Description: as for outcome 8
Time Frame: Day 0 to day 14
Population: Intent to treat. This study had a shared placebo group meaning some participants are included in the analysis for multiple placebo comparison groups. Per master protocol design patients randomized to placebo had the potential to be included in the analyses for infliximab, abatacept, and cenicriviroc based on their eligibility. Therefore, the counts of participants will be higher than the number of participants enrolled. Missing data: Infliximab arms 49, Abatacept arms 57, CVC arms 27.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 506 | 506 | 493 | 499 | 350 | 346
units on a scale | 6.0 (2.4124) | 5.7 (2.5183) | 5.8 (2.3911) | 5.7 (2.5152) | 5.7 (2.4998) | 5.8 (2.4102)
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; p = 0.0903, t-test, 2 sided; Mean Difference (Net) = 0.26, 95% CI 2-sided [-0.04 to 0.57]
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; p = 0.3480, t-test, 2 sided; Mean Difference (Net) = 0.15, 95% CI 2-sided [-0.16 to 0.45]
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; p = 0.6984, t-test, 2 sided; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.44 to 0.29]

13. Secondary Outcome: Mean Change in the 8-point Ordinal Scale From Day 0 to Day 21
Description: as for outcome 8
Time Frame: Day 0 to day 21
Population: Intent to treat. This study had a shared placebo group meaning some participants are included in the analysis for multiple placebo comparison groups. Per master protocol design patients randomized to placebo had the potential to be included in the analyses for infliximab, abatacept, and cenicriviroc based on their eligibility. Therefore, the counts of participants will be higher than the number of participants enrolled. Missing data: Infliximab arms 57, Abatacept arms 64, CVC arms 35.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 501 | 503 | 489 | 496 | 342 | 346
units on a scale | 6.3 (2.4025) | 6.0 (2.5732) | 6.1 (2.4161) | 5.9 (2.5887) | 5.9 (2.6111) | 6.2 (2.4540)
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; p = 0.0450, t-test, 2 sided; Mean Difference (Net) = 0.32, 95% CI 2-sided [0.01 to 0.62]
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; p = 0.2462, t-test, 2 sided; Mean Difference (Net) = 0.19, 95% CI 2-sided [-0.13 to 0.50]
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; p = 0.2304, t-test, 2 sided; Mean Difference (Net) = -0.23, 95% CI 2-sided [-0.61 to 0.15]

14. Secondary Outcome: Mean Change in the 8-point Ordinal Scale From Day 0 to Day 28
Description: as for outcome 8
Time Frame: Day 0 to day 28
Population: Intent to treat. This study had a shared placebo group meaning some participants are included in the analysis for multiple placebo comparison groups. Missing data: Infliximab arms 65, Abatacept arms 69, CVC arms 41.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 496 | 500 | 487 | 493 | 338 | 344
units on a scale | 6.5 (2.4344) | 6.1 (2.6229) | 6.4 (2.4560) | 6.1 (2.6474) | 6.1 (2.6587) | 6.3 (2.4869)
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; p = 0.0313, t-test, 2 sided; Mean Difference (Net) = 0.35, 95% CI 2-sided [0.03 to 0.66]
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; p = 0.0555, t-test, 2 sided; Mean Difference (Net) = 0.31, 95% CI 2-sided [-0.01 to 0.63]
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; p = 0.2710, t-test, 2 sided; Mean Difference (Net) = -0.22, 95% CI 2-sided [-0.60 to 0.17]

15. Secondary Outcome: Duration (Days) Alive and Free of Supplemental Oxygen
Description: Days alive and free of supplemental oxygen
Time Frame: Day 1 to day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 531 | 530 | 524 | 525 | 360 | 363
days | 16.3 (9.87) | 15.2 (10.21) | 15.7 (9.95) | 15.0 (10.35) | 15.3 (10.07) | 15.8 (9.91)
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; Mean Difference (Net) = 1.0, 95% CI 2-sided [-0.0 to 2.0]
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; Mean Difference (Net) = 0.6, 95% CI 2-sided [-0.5 to 1.6]
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.8 to 0.7]

16. Secondary Outcome: Number of Patients With New Supplemental Oxygen Use
Description: Number of patients with new supplemental oxygen use
Time Frame: Day 1-day 28
Population: Intent to treat in patients who were not taking any supplemental oxygen at baseline. This study had a shared placebo group meaning some participants are included in the analysis for multiple placebo comparison groups. Per master protocol design patients randomized to placebo had the potential to be included in the analyses for infliximab, abatacept, and cenicriviroc based on their eligibility. Therefore, the counts of participants will be higher than the number of participants enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 24 | 20 | 25 | 20 | 16 | 13
Participants | 13 | 5 | 11 | 6 | 4 | 4
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; Difference in percentages = 29.2, 95% CI 2-sided [-0.4 to 53.7]
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; Difference in percentages = 14.0, 95% CI 2-sided [-14.8 to 40.0]
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; Difference in percentages = -5.8, 95% CI 2-sided [-38.7 to 26.6]

17. Secondary Outcome: Duration (Days) Alive and Free of Non-invasive Ventilation/ High Flow Oxygen
Description: Days alive and free of non-invasive ventilation/ high flow oxygen
Time Frame: Day 1 to day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 531 | 530 | 524 | 525 | 360 | 363
days | 20.7 (10.20) | 19.5 (11.02) | 20.3 (10.16) | 19.3 (11.12) | 19.4 (11.02) | 20.1 (10.47)
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; Mean Difference (Net) = 1.2, 95% CI 2-sided [0.2 to 2.3]
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; Mean Difference (Net) = 0.9, 95% CI 2-sided [-0.1 to 2.0]
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; Mean Difference (Net) = -0.7, 95% CI 2-sided [-2.0 to 0.6]

18. Secondary Outcome: Number of Patients With New Non-invasive Ventilation/High Flow Oxygen Use
Description: Number of patients with new non-invasive ventilation/high flow oxygen use
Time Frame: Day 1-day 28
Population: Intent to treat in patients who were not taking any supplemental or non-invasive/high flow oxygen at baseline. Per master protocol design patients randomized to placebo had the potential to be included in the analyses for infliximab, abatacept, and cenicriviroc based on their eligibility. Therefore, the counts of participants will be higher than the number of participants enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 299 | 299 | 301 | 299 | 201 | 204
Participants | 68 | 89 | 81 | 92 | 64 | 67
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; Difference in percentages = -7.0, 95% CI 2-sided [-14.0 to 0.0]
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; Difference in percentages = -3.9, 95% CI 2-sided [-11.1 to 3.4]
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; Difference in percentages = -1.0, 95% CI 2-sided [-10.1 to 8.1]

19. Secondary Outcome: Duration (Days) Alive and Free of Invasive Mechanical Ventilation or ECMO
Description: Days alive and free of invasive mechanical ventilation or ECMO
Time Frame: Day 1 to day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 531 | 530 | 524 | 525 | 360 | 363
days | 23.4 (8.96) | 22.6 (9.75) | 23.4 (9.16) | 22.6 (9.72) | 22.4 (9.95) | 23.2 (9.17)
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; Mean Difference (Net) = 0.9, 95% CI 2-sided [-0.1 to 1.8]
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; Mean Difference (Net) = 0.7, 95% CI 2-sided [-0.3 to 1.7]
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; Mean Difference (Net) = -0.8, 95% CI 2-sided [-2.0 to 0.4]

20. Secondary Outcome: Number of Patients With New Mechanical Ventilation or ECMO Use
Description: Number of patients with new mechanical ventilation or ECMO use
Time Frame: Day 1 to day 28
Population: Intent to treat in patients that were not receiving ECMO at baseline. This study had a shared placebo group meaning some participants are included in the analysis for multiple placebo comparison groups. Per master protocol design patients randomized to placebo had the potential to included in the analyses for infliximab, abatacept, and cenicriviroc based on their eligibility. Therefore, the counts of participants will be higher than the number of participants enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 473 | 477 | 476 | 474 | 331 | 332
Participants | 70 | 76 | 71 | 77 | 62 | 55
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; Difference in percentages = -1.1, 95% CI 2-sided [-5.7 to 3.5]
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; Difference in percentages = -1.3, 95% CI 2-sided [-6.0 to 3.3]
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; Difference in percentages = 2.2, 95% CI 2-sided [-3.7 to 8.0]

21. Secondary Outcome: Duration (Days) Alive and Out of the Hospital
Description: Days alive and out of the hospital
Time Frame: Through day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 531 | 530 | 524 | 525 | 360 | 363
days | 14.7 (9.42) | 13.8 (9.74) | 14.1 (9.75) | 13.7 (9.86) | 14.2 (9.56) | 14.3 (9.56)
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; Mean Difference (Net) = 1.0, 95% CI 2-sided [-0.0 to 2.0]
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; Mean Difference (Net) = 0.4, 95% CI 2-sided [-0.7 to 1.4]
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; Mean Difference (Net) = -0.1, 95% CI 2-sided [-1.3 to 1.1]

22. Secondary Outcome: Number of Patients With SAEs Through Day 28
Description: Cumulative Incidence of SAEs through day 28
Time Frame: Day 28
Population: Modified intent to treat. This study had a shared placebo group meaning some participants are included in the analysis for multiple placebo comparison groups. Per master protocol design patients randomized to placebo had the potential to be included in the analyses for infliximab, abatacept, and cenicriviroc based on their eligibility. Therefore, the counts of participants will be higher than the number of participants enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 517 | 516 | 509 | 510 | 355 | 354
Participants | 112 | 124 | 116 | 131 | 95 | 80
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; p = 0.3169, Log Rank; Hazard Ratio (HR) = 0.878, 95% CI 2-sided [0.680 to 1.133]
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; p = 0.2480, Log Rank; Hazard Ratio (HR) = 0.863, 95% CI 2-sided [0.672 to 1.108]
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; p = 0.2490, Log Rank; Hazard Ratio (HR) = 1.191, 95% CI 2-sided [0.885 to 1.604]

23. Secondary Outcome: Number of Patients With Grade 3 and 4 Adverse Events
Description: Cumulative incidence of adverse events of grade 3 and 4
Time Frame: Day 28
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 517 | 516 | 509 | 510 | 355 | 354
Participants | 137 | 126 | 124 | 132 | 101 | 94
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; p = 0.5175, Log Rank; Hazard Ratio (HR) = 1.083, 95% CI 2-sided [0.850 to 1.380]
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; p = 0.5216, Log Rank; Hazard Ratio (HR) = 0.923, 95% CI 2-sided [0.722 to 1.179]
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; p = 0.6135, Log Rank; Hazard Ratio (HR) = 1.075, 95% CI 2-sided [0.812 to 1.424]

24. Secondary Outcome: Number of Patients With Adverse Events Leading to Dose Modification
Description: Number of patients with adverse events (serious and non serious) leading to dose modification
Time Frame: Day 1-28
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
Number analyzed (Participants) | 517 | 516 | 509 | 510 | 355 | 354
Participants | 4 | 7 | 4 | 7 | 34 | 7
Statistical Analysis 1: Comparison: Standard of Care + Infliximab vs Standard of Care + Infliximab Matching Placebo; Test type: Superiority; p = 0.3628, Log Rank; Hazard Ratio (HR) = 0.565, 95% CI 2-sided [0.165 to 1.931]
Statistical Analysis 2: Comparison: Standard of Care + Abatacept vs Standard of Care + Abatacept Matching Placebo; Test type: Superiority; p = 0.3701, Log Rank; Hazard Ratio (HR) = 0.570, 95% CI 2-sided [0.167 to 1.948]
Statistical Analysis 3: Comparison: Standard of Care + Cenicriviroc vs Standard of Care + Cenicriviroc Matching Placebo; Test type: Superiority; p = 0.0001, Log Rank; Hazard Ratio (HR) = 4.988, 95% CI 2-sided [2.211 to 11.251]

ADVERSE EVENTS:
Time Frame: Day 1-60
Description: Adverse events were collected on a modified intent to treat population during hospitalization days and at time of outpatient visits. All-cause mortality was collected on intent to treat population.
  This study had a shared placebo group meaning some participants are included in the analysis for multiple placebo comparison groups.
Groups:
- Standard of Care + Infliximab Matching Placebo: infliximab matching placebo (single dose IV 5mg/kg given on day 1)
  Remdesivir: Standard of Care
- Standard of Care + Abatacept Matching Placebo: abatacept matching placebo (single dose IV 10 mg/kg up to 1,000 mg given on day 1)
  Remdesivir: Standard of Care
- Standard of Care + Cenicriviroc: cenicriviroc [tablet, Day 1/Loading Dose: 450 mg (300mg morning and 150mg evening) Day 2 - 29/Maintenance Dose: 300 mg (150 mg BID) through Day 29].
  cenicriviroc: study drug
  Remdesivir: Standard of Care
  cenicriviroc (closed to enrollment as of 3-Sep-2021): study drug
- Standard of Care + Cenicriviroc Matching Placebo: cenicriviroc matching placebo [tablet, Day 1/Loading Dose: 2 tabs in morning and 1 evening Day 2 - 29/Maintenance Dose: BID through Day 29].
  Remdesivir: Standard of Care
Arm/Group | Standard of Care + Infliximab | Standard of Care + Infliximab Matching Placebo | Standard of Care + Abatacept | Standard of Care + Abatacept Matching Placebo | Standard of Care + Cenicriviroc | Standard of Care + Cenicriviroc Matching Placebo
All-Cause Mortality (participants affected / at risk) | 65/531 | 85/530 | 74/524 | 87/525 | 64/360 | 49/363
Serious Adverse Events (participants affected / at risk) | 125/517 | 130/516 | 128/509 | 136/510 | 102/355 | 84/354
Other Adverse Events (participants affected / at risk) | 18/517 | 18/516 | 24/509 | 18/510 | 13/355 | 13/354
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care + Infliximab (N=517) | Standard of Care + Infliximab Matching Placebo (N=516) | Standard of Care + Abatacept (N=509) | Standard of Care + Abatacept Matching Placebo (N=510) | Standard of Care + Cenicriviroc (N=355) | Standard of Care + Cenicriviroc Matching Placebo (N=354)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 11 | 5 | 11 | 8 | 7
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 36 | 36 | 35 | 39 | 37 | 30
Pneumonia (Infections and infestations) | 8 | 13 | 16 | 11 | 14 | 6
Acute kidney injury (Renal and urinary disorders) | 11 | 9 | 8 | 8 | 7 | 4
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 32 | 29 | 23 | 32 | 21 | 17
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 5 | 11 | 7 | 13 | 5 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 3 | 2 | 5 | 0
Septic shock (Infections and infestations) | 9 | 7 | 14 | 8 | 6 | 5
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 3 | 7 | 3 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 3 | 2 | 4 | 0
Pneumonia bacterial (Infections and infestations) | 5 | 5 | 3 | 5 | 3 | 3
Sepsis (Infections and infestations) | 5 | 3 | 5 | 3 | 2 | 2
Deep Vein Thrombosis (Vascular disorders) | 5 | 3 | 1 | 3 | 0 | 3
Cardiac arrest (Cardiac disorders) | 7 | 2 | 6 | 2 | 6 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care + Infliximab (N=517) | Standard of Care + Infliximab Matching Placebo (N=516) | Standard of Care + Abatacept (N=509) | Standard of Care + Abatacept Matching Placebo (N=510) | Standard of Care + Cenicriviroc (N=355) | Standard of Care + Cenicriviroc Matching Placebo (N=354)
Pneumonia (Infections and infestations) | 18 | 18 | 24 | 18 | 13 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Study Protocol (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT04593940/Prot_001.pdf
  • Statistical Analysis Plan (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT04593940/SAP_002.pdf
  • Informed Consent Form (2020-12-31): https://cdn.clinicaltrials.gov/large-docs/40/NCT04593940/ICF_000.pdf